CLINICAL TRIAL: NCT03937011
Title: A Prospective, Multicenter, Multispecialty Evaluation of STRATAFIX™ Spiral PDS™ Plus Knotless Tissue Control Devices in Robotic Procedures
Brief Title: Post-Market Clinical Follow-Up of STRATAFIX™ Spiral PDS™ PLUS
Status: Completed | Type: Observational
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ESC_2018_02
Record Dates: First submitted 2019-04-26; First posted 2019-05-03 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Bariatric - Sleeve Gastrectomy Staple Line Reinforcement; Gynecology - Vaginal Cuff Closure
Keywords: STRATAFIX SPIRAL PDS PLUS, ROBOTIC SUTURING,

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Stratafix Arm: The single study arm would comprise of two different specialties in Robotic surgical procedures: Bariatric Sleeve gastrectomy (Staple line reinforcement) and Hysterectomy (Vaginal cuff closure).
  Interventions: Device: Robotic Suturing of gastric sleeve oversew and vaginal cuff closure

INTERVENTIONS:
Device: Robotic Suturing of gastric sleeve oversew and vaginal cuff closure — 1. Robotic Bariatric Sleeve gastrectomy
  2. Robotic Hysterectomy with or without oophorectomy;

SUMMARY:
This single-arm, prospective, observational multicenter study will collect clinical data in a post-market setting across two different specialties in Robotic surgical procedures: Bariatric Sleeve gastrectomy (Staple line reinforcement) and Hysterectomy (Vaginal cuff closure). Investigators will perform the procedure using SFX Spiral PDS Plus in compliance with their standard surgical approach and the IFU.

ELIGIBILITY:
Inclusion:

1. Elect to have a Robotic Bariatric Sleeve Gastrectomy or Robotic Total Hysterectomy where STRATAFIX™ Spiral PDS™ Plus device is used for staple line re-enforcement or vaginal cuff closure, respectively
2. Are willing and able to give consent and comply with all study-related evaluations and treatment scheduled
3. Subjects are ≥ 18 years of age

Exclusion:

1. Physical or psychological condition which would impair study participation or are unwilling or unable to participate in all required study visits
2. Any pre-operative or intra-operative findings identified by the surgeon that may preclude the use of study product
3. Enrolled in a concurrent clinical study (drug/device) that might affect current study primary or secondary endpoints
4. Allergic to poly (p-dioxanon), IRGACARE®* MP (triclosan) or D&C Violet No. 2 colorant
5. Pregnant or lactating female subjects as confirmed prior to the procedure
6. Subjects undergoing radical hysterectomy (Type B, C and D) according to Querleu & Morrow classification or gastric sleeve revision surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects ≥ 18 years who are undergoing elective/non-emergent gastric or gynecological procedures robotically
Sampling Method: Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with no bleeding or mild bleeding (defined as success) at the completion of the suturing at the organ layer (vaginal cuff closure or gastric staple line reinforcement using STRATAFIX™ Spiral PDS™ Plus). | Intra-op assessment (During Surgery; after suturing of the target tissue, Day of surgery)
  The bleeding grade assessment used for the primary endpoint will be made right after the suturing is completed. Any re-bleeding after the initial assessment (just before the removal of the optics and trocars) from the suture line after this assessment will be considered a failure for the primary performance endpoint.

SECONDARY OUTCOMES:
Qualitative Assessment of Suture Handling | Intra-op (at surgery, after suturing of the target tissue layer, Day of surgery)
  Suture breakage, correction suture used, reinforcement suture used, needle penetration, size, attachment; all rated 1-5
Time to Closure (in minutes/seconds) | Intra-op (during suturing of the target tissue, Day of surgery)
  The time to closure is defined as time in minutes and seconds between placement of the first suture throw in the target tissue to the completion of closure of that layer. The time in minutes and seconds will be captured as per operating room procedure.
Overall procedure time (first incision to skin closure) | Intra-op (during the surgery, Day of surgery)
  Overall time is calculated as first incision to skin closure
Length of stay in hours | Post-Operative up to 48 hrs
  Time from admission to discharge
Estimated intra-operative blood loss per institutional standard of care and incidence of subjects requiring blood transfusion | Intra-Op (during the surgery, Day of surgery)
  Blood loss calculated as per the standard of care of each institution
Intra-operative leak test in bariatric procedure as per institutional standard of care, if any | Intra-op (during Surgery; Day of surgery)
  Leak test for sleeve gastrectomy patient as per institution standard
Post-operative male/female dyspareunia related to sutures (total hysterectomy subjects) | 90 days post-operative (+/- 30 days), 180 days post-operative (+/- 30 days)
  Dyspareunia here is defined as painful sexual intercourse due to the sutures
Incisional site physical assessment:is suture palpable, suture line intact, or tender (all rated yes/no) | 14 days post-perative 90 days post-operative (+/- 30 days), 180 days post-operative (+/- 30 days)
  Incisional site will be assessed for hysterectomy subjects to see if the suture is palpable suture, tender or intact at the target site
Abnormal vaginal discharge (total hysterectomy subjects) | 14 days post-perative 90 days post-operative (+/- 30 days), 180 days post-operative (+/- 30 days)
  Hysterectomy patients will be assessed for any abnormal vaginal discharge if any.
C-SATS GEARS score | Intra-op (during the surgery, Day of surgery)
  Global Evaluative Assessment of Robotic Skills (GEARS). Its a validated assessment tool for grading overall technical proficiency for robotic surgery. GEARS measures manual dexterity and fluidity of motion and does not define surgical or clinical judgement. The scales are Depth perception, Bimanual dexterity, efficiency, force sensitivity and robotic control.Each scale is scored 1 - 5, which means the total score could range from 5 - 25.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (4):
  - Baptist Health South Florida, Miami, Florida
  - Albany Medical, Albany, New York
  - Mt. Sinai, New York, New York
  - Lenox Hill hospital, New York, New York
- Germany (2):
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - Klinuk fur Allgemelne, Viszeral-ThoraxTransplantations- und Kinderchirurgie, Kiel
- Italy (2):
  - University of Naples, Naples
  - University Pisa, Pisa

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu